CLINICAL TRIAL: NCT01744236
Title: A Phase IV, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Assess the Effect of 12-week Treatment With the Glucagon-like Peptide-1 Receptor Agonist (GLP-1RA) Liraglutide or Dipeptidyl Peptidase-4 Inhibitor (DPP-4i) Sitagliptin on the Cardiovascular, Renal and Gastrointestinal System in Insulin-naïve Patients With Type 2 Diabetes (T2DM).
Brief Title: SAFEGUARD: Pleiotropic Effects of Incretin Based Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: EU FP7: SAFEGUARD consortium (Unknown)
Responsible Party: Principal Investigator, M.H.H. Kramer, Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DC2012SAFE001; U1111-1130-8248 (Other: WHO Universal Trial Number); 2012-003256-36 (EudraCT Number)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1 Receptor Agonists, DPP-4 inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate; Exenatide; omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Liraglutide (main study, long-term intervention) (Experimental): This arm (n=20) will receive liraglutide 1.8mg and sitagliptin-placebo during 12 weeks
  Interventions: Drug: Liraglutide; Drug: Sitagliptin placebo
- Sitagliptin (main study, long-term intervention) (Experimental): This arm (n=20) will receive sitagliptin 100mg and liraglutide-placebo during 12 weeks
  Interventions: Drug: Sitagliptin; Drug: Liraglutide placebo
- Placebo (main study, long-term intervention) (Placebo Comparator): This arm (n=20) will receive liraglutide-placebo and sitagliptin-placebo during 12 weeks
  Interventions: Drug: Liraglutide placebo; Drug: Sitagliptin placebo
- Exenatide (main study, acute intervention) (Experimental): Prior to the 12-week intervention study, a GLP-1 receptor agonist (exenatide) will be administered intravenously (n=30).
  Interventions: Drug: Exenatide
- Placebo (main study, acute intervention) (Placebo Comparator): Prior to the 12-week intervention study, placebo will be administered intravenously (n=30).
  Interventions: Drug: Exenatide placebo
- Acute MRI intervention study (Other): In a subset of 12 patients with type 2 diabetes, a crossover trial with acute infusion of exenatide and placebo is performed. This is done prior to the 12-week intervention study.
  Interventions: Drug: Exenatide; Drug: Exenatide placebo
- Pilot-study (Other): In 10 healthy obese subjects, a crossover trial with acute infusion of exenatide, placebo and L-NMMA is performed.
  Interventions: Drug: Exenatide; Drug: Exenatide placebo; Drug: L-NMMA

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be started with a titration period of 2 weeks (week 1: 0.6mg once daily and week 2: 1.2mg once daily). If liraglutide is well tolerated it will be continued for 10 more weeks in a dosage of 1.8mg once daily.
  Arms: Liraglutide (main study, long-term intervention)
Drug: Sitagliptin — Sitagliptin 100mg will be given once daily for 12 weeks.
  Arms: Sitagliptin (main study, long-term intervention)
Drug: Exenatide — Exenatide will be administered intravenously with a loading dose of 50ng/min for 30 minutes, followed by a maintenance dose of 25ng/min during the rest of the tests
  Arms: Acute MRI intervention study; Exenatide (main study, acute intervention); Pilot-study
Drug: Liraglutide placebo — Liraglutide-placebo will be started with a titration period of 2 weeks (week 1: 0.6mg once daily and week 2: 1.2mg once daily). It will be continued for 10 more weeks in a dosage of 1.8mg once daily.
  Arms: Placebo (main study, long-term intervention); Sitagliptin (main study, long-term intervention)
Drug: Sitagliptin placebo — Sitagliptin-placebo be given once daily for 12 weeks.
  Arms: Liraglutide (main study, long-term intervention); Placebo (main study, long-term intervention)
Drug: Exenatide placebo — Exenatide-placebo (saline) will be administered intravenously
  Arms: Acute MRI intervention study; Pilot-study; Placebo (main study, acute intervention)
Drug: L-NMMA
  Arms: Pilot-study

SUMMARY:
The aim of this study is to detail the (mechanisms underlying the) actions of the GLP-1 receptor agonists and DPP-4 inhibitors on the cardiovascular, renal and gastrointestinal systems in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
GLP-1 receptors are present in most organ systems of the human body, and pharmacological interventions enhancing GLP-1 activity may influence the function of these organs. The use of GLP-1 receptor agonists (GLP-1RA) and DPP-4 inhibitors (DPP-4i) has been associated with an increased heart rate, acute pancreatitis and acute renal failure. To date, studies in humans detailing the effects of these drugs on these organ systems, biological processes and underlying mechanisms, which could explain these associations, are lacking.

Therefore, as part of the EU-FP7 SAFEGUARD program, the present study will aim to detail the (mechanisms underlying the) actions of GLP-1RA and DPP-4i on the cardiovascular, renal and gastrointestinal system in healthy obese subjects and patients with T2DM.

In the main study, sixty patients with type 2 diabetes will undergo two interventions within the same protocol in order to assess changes in the outcome parameters:

* acute study = acute infusion with exenatide or placebo (to assess the cardiovascular and renal effects)
* long-term study = 12 weeks of treatment with liraglutide, sitagliptin or placebo (to assess the cardiovascular, renal and gastrointestinal effects)

In a substudy (termed 'acute MRI study'), twelve patients with type 2 diabetes will undergo an additional acute intervention study with exenatide (to assess the pancreatic effects)

In a substudy (termed 'pilot-study'), ten healthy obese subjects will undergo a similar acute study like the patients with type 2 diabetes (to assess the cardiovascular and renal effects). Moreover, in these healthy subjects, the effects of exenatide during L-NMMA infusion will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 75 years.
* Females must be post-menopausal (no menses >1 year).
* Type 2 diabetes (HbA1c 6.5-9% DCCT or 48-75 mmol/mol IFCC), who are being treated with a stable dose of oral antihyperglycemic agents (either metformin alone, SU alone or a combination of metformin and SU) for at least 3 months prior to inclusion.
* BMI 25 - 40 kg/m2
* Caucasian
* Signed informed consent

Exclusion Criteria:

* GFR < 60 mL/min/1.73m2
* Current / chronic use of the following medication: thiazolidinediones, GLP-1RA, DPP-4i, glucocorticoids, NSAIDs, insulin, antimicrobial agents, chemotherapeutics or immune suppressants. Subjects on diuretics will only be excluded when these drugs (e.g. hydrochlorothiazide) cannot be stopped for the duration of the study.
* History of or actual pancreatic disease or impaired pancreatic exocrine function
* Active liver disease
* History of or actual malignancy (with the exception of basal cell carcinoma)
* Current urinary tract infection and active nephritis
* Recent (<6 months) history of cardiovascular disease, including acute coronary syndrome, stroke, transient ischemic neurologic disorder or chronic heart failure (New York Heart Association grade II-IV)
* Current atrial fibrillation
* Chronic infectious or auto-immune disease
* Substance and/or alcohol abuse
* History of allergy/hypersensitivity to any of the test agents
* Complaints compatible with or established gastroparesis and/or neurogenic bladder
* Any condition that has been recognized as a contra-indication for the use of GLP-1RA and DPP-4i, as listed in the respective SPCs
* History of or actual (severe) mental illness
* Inability to understand the study protocol and/or inability to give informed consent
* History of claustrophobia or presence of metal objects/implants (because of MRI protocol)

For the preceding Pilot study, we will include:

* Males
* Age between 18 and 50 years
* BMI 25 - 40 kg/m2
* Caucasian

The exclusion criteria for the preceding pilot study are similar to the exclusion criteria of the main study, with the additions of:

* Subjects with a fasting plasma glucose ≥5.6 mmol/L, a 2-hour glucose of ≥7.8 mmol/L after a 75-grams oral glucose tolerance test, or a HbA1c of ≥6.5%
* Subjects using any kind of medication

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline following infusion of GLP-1RA (acute effects) and the changes from baseline following 12-week treatment with GLP-1RA or DPP-4i (long-term effects) on resting heart rate variability, as derived from electrocardiographic measurements. | 12 weeks
Changes from baseline following infusion of GLP-1RA (acute effects) and the changes from baseline following 12-week treatment with GLP-1RA or DPP-4i (long-term effects) on Glomerular Filtration Rate, measured by the inulin-clearance technique. | 12 weeks
Changes from baseline following 12-week treatment with GLP-1RA or DPP-4i (long-term effects) on pancreatic exocrine function, measured as fecal Elastase-1. | 12 weeks

SECONDARY OUTCOMES:
Changes from baseline following infusion of GLP-1RA (acute effects) and the changes from baseline following 12-week treatment with GLP-1RA or DPP-4i (long-term effects) on the following cardiovascular parameters: | 12 weeks
  * Blood pressure and heart rate
  * Hemodynamic variables (blood pressure, heart rate, stroke volume, cardiac output/-index/-contractility, systemic vascular resistance) derived from non-invasive beat-to-beat finger blood pressure measurements
  * Cardiac autonomic nervous system function
  * Microvascular function and vasomotion
  * Arterial stiffness
  * Lipid spectrum
  * Glycemic variables (HbA1c, fasting and postprandial glucose)
  * Body anthropometrics: body weight, height, BMI and waist circumference
  * Body fat content
Changes from baseline following infusion of GLP-1RA (acute effects) and the changes from baseline following 12-week treatment with GLP-1RA or DPP-4i (long-term effects) on the following renal parameters: | 12 weeks
  * Effective renal plasma flow (ERPF)
  * Renal tubular function
  * Renal damage, measured by urine biomarkers
Changes from baseline following infusion of GLP-1RA (acute effects*) and changes from baseline following 12-week treatment with GLP-1RA or DPP-4i (long-term effects) on the following gastrointestinal parameters: | 12 weeks
  * Pancreatic exocrine function (* In the acute intervention only exocrine pancreatic function is assessed)
  * Pancreatic structure
  * Pancreatic enzymes
  * Gallbladder emptying speed
  * Liver enzymes
  * Hepatic structure/steatosis
  * Gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: M.H.H. Kramer, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Smits MM, Fluitman KS, Herrema H, Davids M, Kramer MHH, Groen AK, Belzer C, de Vos WM, Cahen DL, Nieuwdorp M, van Raalte DH. Liraglutide and sitagliptin have no effect on intestinal microbiota composition: A 12-week randomized placebo-controlled trial in adults with type 2 diabetes. Diabetes Metab. 2021 Sep;47(5):101223. doi: 10.1016/j.diabet.2021.101223. Epub 2021 Jan 8. PMID 33429063
- [Derived] Smits MM, Tonneijck L, Muskiet MH, Kramer MH, Pouwels PJ, Pieters-van den Bos IC, Hoekstra T, Diamant M, van Raalte DH, Cahen DL. Twelve week liraglutide or sitagliptin does not affect hepatic fat in type 2 diabetes: a randomised placebo-controlled trial. Diabetologia. 2016 Dec;59(12):2588-2593. doi: 10.1007/s00125-016-4100-7. Epub 2016 Sep 15. PMID 27627981
- [Derived] Tonneijck L, Smits MM, Muskiet MH, Hoekstra T, Kramer MH, Danser AH, Ter Wee PM, Diamant M, Joles JA, van Raalte DH. Renal Effects of DPP-4 Inhibitor Sitagliptin or GLP-1 Receptor Agonist Liraglutide in Overweight Patients With Type 2 Diabetes: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Trial. Diabetes Care. 2016 Nov;39(11):2042-2050. doi: 10.2337/dc16-1371. Epub 2016 Sep 1. PMID 27585605
- [Derived] Smits MM, Tonneijck L, Muskiet MH, Hoekstra T, Kramer MH, Diamant M, Nieuwdorp M, Groen AK, Cahen DL, van Raalte DH. Biliary effects of liraglutide and sitagliptin, a 12-week randomized placebo-controlled trial in type 2 diabetes patients. Diabetes Obes Metab. 2016 Dec;18(12):1217-1225. doi: 10.1111/dom.12748. Epub 2016 Aug 30. PMID 27451030
- [Derived] Tonneijck L, Smits MM, Muskiet MHA, Hoekstra T, Kramer MHH, Danser AHJ, Diamant M, Joles JA, van Raalte DH. Acute renal effects of the GLP-1 receptor agonist exenatide in overweight type 2 diabetes patients: a randomised, double-blind, placebo-controlled trial. Diabetologia. 2016 Jul;59(7):1412-1421. doi: 10.1007/s00125-016-3938-z. Epub 2016 Apr 1. PMID 27038451
- [Derived] Smits MM, Tonneijck L, Muskiet MH, Hoekstra T, Kramer MH, Pieters IC, Cahen DL, Diamant M, van Raalte DH. Cardiovascular, renal and gastrointestinal effects of incretin-based therapies: an acute and 12-week randomised, double-blind, placebo-controlled, mechanistic intervention trial in type 2 diabetes. BMJ Open. 2015 Nov 19;5(11):e009579. doi: 10.1136/bmjopen-2015-009579. PMID 26586327
- See also: The website of the European project SAFEGUARD — http://www.safeguard-diabetes.org/